CLINICAL TRIAL: NCT02101398
Title: Etude de l'Effet de Stimulations transcrâniennes en Courant Continu (tDCS) Sur Les Performances en dénomination Chez le Sujet Aphasique à Moins d'un an de Son Accident Vasculaire cérébral : Comparaison de 5 Configurations de Stimulation
Brief Title: Study of the Effect of Transcranial Stimulations in Aphasic Subject Within a Year of Their Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low inclusion rate
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: C12-09; 2013-A00989-36 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-03-21; First posted 2014-04-02 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2021-08

CONDITIONS: Aphasia; Stroke
Keywords: tDCS; Stroke; Aphasia; Naming
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- F7A (Experimental): Anodal electrode set on the left Broca's area and cathodal electrode set on its right homologue. Active stimulation.
  Interventions: Device: eldith DC-stimulator, configuration F7A
- F7C (Experimental): Cathodal electrode set on the left Broca's area and anodal electrode set on its right homologue. Active stimulation.
  Interventions: Device: eldith DC-stimulator, configuration F7C
- T5A (Experimental): Anodal electrode set on the left Wernicke's area and cathodal electrode set on its right homologue. Active stimulation.
  Interventions: Device: eldith DC-stimulator, configuration T5A
- T5C (Experimental): Cathodal electrode set on the left Wernicke's area and anodal electrode set on its right homologue. Active stimulation.
  Interventions: Device: eldith DC-stimulator, configuration T5C
- Sham (Sham Comparator): Electrodes set on the left Broca's area and its right homologue or electrodes set on the left Wernicke's area and its right homologue, but no stimulation will be delivered.
  Interventions: Device: eldith DC-stimulator, configuration Sham

INTERVENTIONS:
Device: eldith DC-stimulator, configuration F7A — tDCS will be delivered during a 20 minutes speech-language therapy session
  Arms: F7A
Device: eldith DC-stimulator, configuration F7C — tDCS will be delivered during a 20 minutes speech-language therapy session
  Arms: F7C
Device: eldith DC-stimulator, configuration T5A — tDCS will be delivered during a 20 minutes speech-language therapy session
  Arms: T5A
Device: eldith DC-stimulator, configuration T5C — tDCS will be delivered during a 20 minutes speech-language therapy session
  Arms: T5C
Device: eldith DC-stimulator, configuration Sham — Sham tDCS will be delivered during a 20 minutes speech-language therapy session
  Arms: Sham

SUMMARY:
The aim of this work is to study the effect of transcranial direct current stimulation combined with naming therapy in acute and post-acute stroke comparing four bihemispheric positioning electrodes to a sham condition.

DETAILED DESCRIPTION:
TDCS have shown a positive effect on clinical outcome in naming treatment in aphasic subjects however some aspects as the positioning of the electrodes on the head are still unclear. That is why we compare the effects of four different positionings of the electrodes (two anterior over Broca's area and its homologue and two posterior over Wernicke's area and its homologue) to a sham stimulation in order to observe if a more important effect of one or another positioning could be found.

ELIGIBILITY:
Inclusion Criteria:

* man or woman of 18 years and older
* aphasic patient following a first left hemispheric stroke
* BDAE 3.0 aphasia score > or = to 1
* stroke within 3 to 12 months before inclusion in the study
* mother tongue = French
* right handedness
* signed informed consent

Exclusion Criteria:

* history of other neurologic pathologies
* epileptic seizure within 2 months before inclusion
* dementia
* bilingual patient (2 mother tongues)
* history of cranial surgery
* presence of intracerebral metallic material
* unauthorized molecules at inclusion : sulpiride, rivastigmine, dextromethorphan, carbamazepine, flunarizine, levodopa
* pregnant, parturient or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of improvement of picture naming | Before stimulation and immediately after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD, Principal Investigator — Hôpital Raymond Poincaré
Locations (1):
- Hôpital Raymond Poincaré, Garches, France